CLINICAL TRIAL: NCT02499003
Title: The GOAL Trial: Rescue Treatment With the Monoclonal Anti CD20-antibody Obinutuzumab (GA101) in Combination With Pixantrone for the Treatment of Patients With Relapsed Aggressive B-cell Lymphoma
Brief Title: GOAL: GA101 Plus Pixantrone for Relapsed Aggressive Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Roche Pharma AG (Industry); Servier (Industry)
Responsible Party: Principal Investigator, Georg Hess, MD, Principle Ivestigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETN-1 GOAL; 2014-004780-21 (EudraCT Number); ML29498 (Other: Roche trial code)
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Diffuse large B-cell lymphoma; Follicular lymphoma; Transformed indolent lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — obinutuzumab; pixantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Obinutuzumab and Pixantrone (Experimental): Obinutuzumab: 1000 mg flat dose on day 1, 8, 15 of cycle one and day 1 of subsequent cycles Pixantrone: 50 mg/m² Pixantrone on day 1,8,15 of each 28 d cycle
  Interventions: Drug: Obinutuzumab and Pixantrone

INTERVENTIONS:
Drug: Obinutuzumab and Pixantrone — Obinutuzumab: 1000 mg flat dose on day 1, 8, 15 of cycle one and day 1 of subsequent cycles, Pixantrone: 50 mg/m² Pixantrone on day 1,8,15 of each 28 d cycle
  Other Names: GA101 /Gazyvaro; Pixuvri

SUMMARY:
The purpose of this study is to evaluate the overall response rate of Obinutuzumab (GA101) in combination with Pixantrone in patients with relapsed aggressive B-cell lymphoma. 70 patients with diffuse large B-cell lymphoma, follicular lymphoma grade IIIB or transformed indolent lymphoma will receive up to 6 cycles of the described combination regimen. Follow up visits are scheduled for up to 3 years.

DETAILED DESCRIPTION:
In patients with multiple relapsed aggressive lymphoma or refractory lymphoma life expectancy is short. Without potent treatment options the remaining life span can be measured in weeks to a few months.

Recently, an increasing number of reports have shown that either single agent use or the incorporation of potentially more potent agents or new approaches aiming at the inhibition of lymphoma specific pathways may help to overcome the current stagnation in the improvement of first and second line therapies. Surprisingly, little efforts have been undertaken to identify optimal standard dose backbone regimens based on currently available and novel drugs, which ideally would combine activity with reasonable safety and tolerability which allows the addition of targeted drugs in the future. Therefore this trial aims to test prospectively one potential combination to evaluate its potency in patients not suitable for intensive treatment.

Obinutuzumab is an anti-CD20 monoclonal antibody which has shown clinical efficacy even in patients failing Rituximab pre-treatment and therefore is an attractive combination partner within chemo-immunotherapy regimen. Pixantrone belongs to the most potent class of cytostatic drugs for the treatment of lymphoma. Given the proven efficacy of both drugs in relapsed aggressive lymphoma as well as the side effect profiles of both drugs, combination treatment seems sufficiently safe and promises significant efficacy.

This is a multicenter, prospective, open-label, non-randomized trial to evaluate the overall response rate of Obinutuzumab (GA101) in combination with Pixantrone in patients with relapsed aggressive B-cell lymphoma. The trial consists of a 28-days screening period, a treatment-period of up to 6 cycles of the combination regiment, including an interim staging prior to cycle 4 and an end of treatment visit 4-6 weeks after the last study-medication application. The response to treatment is measured by results of computer tomography (CT) after cycle 6 or at the individual end of treatment. Structured follow up visits are scheduled for 2 years, afterwards patients will be followed for survival and progression via a simplified survey until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Histologically proven diagnosis of diffuse large cell B-cell lymphoma (DLBCL), follicular lymphoma (FL) IIIB or transformed indolent lymphoma according to the World Health Organization classification (central pathology review)
* Relapsed disease
* Eastern Cooperative Oncology Group (ECOG) performance Status ≤2, unless tumor associated
* Adequate cardiac reserve: Serum Troponin level must be consistent with no significant acute or chronic myocardial damage and there should be no evidence of symptomatic disease
* No curative option available
* At least 1 measurable tumor mass (>1.5 cm x >1.0 cm) or bone marrow infiltration
* Adequate bone marrow (BM) reserve: Platelets of at least 100.000/µl (in case of extensive BM-infiltration 75.000/µl may be acceptable after discussion with the coordinating investigator), absolute neutrophil count of at least 1000/µl. Adequate hepatic and renal function: Alanine aminotransferase <2.5 x upper limit of normal (ULN); Aspartate aminotransferase <2.5 x ULN, total bilirubin <1.5 x ULN
* No active Hepatitis B or C or HIV-infection
* Measured or calculated creatinine clearance >30 mL/min
* Fresh tumor biopsy or archived tissue available
* Ability of patients to understand nature, importance and individual consequences of clinical trial.
* Signed informed consent
* Women post-menopausal for more than two years can participate in the trial. Women with childbearing potential can only participate, if they are surgically sterile or a negative pregnancy test (serum or urine) is available before trial and they are willing to practice a highly effective and medically accepted contraception method during trial and for a period of 18 months post-treatment. Reliable contraception comprises systematic contraceptives (oral, implant, injection) or diaphragm / condoms / intrauterine devices (IUP) with spermicide.
* Male patients are advised to use contraceptive methods (preferably barrier) during treatment and for a period of 6 months post-treatment

Exclusion Criteria:

* Lymphoma other than DLBCL, FL IIIB, transformed indolent Non-Hodgkin's lymphoma (NHL)
* Central nervous System (CNS) involvement (brain MRI (Magnetic resonance Imaging) is required only in cases of clinically suspicious involvement)
* Pregnant or breast-feeding women
* Severe concomitant disease (e.g. uncontrolled arterial hypertension, heart failure (NYHA III-IV), uncontrolled diabetes mellitus, pulmonary fibrosis, uncontrolled hyperlipoproteinaemia)
* Myocardial infarction within the last 6 months
* Active uncontrolled infections including HIV-positivity, active Hepatitis B or C
* Vaccination with live vaccine within last 4 weeks
* Mental status precluding patient's compliance
* Known CD20 negativity
* Diagnosed or treated for a malignancy other than NHL except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, Ductal Carcinoma in Situ (DCIS) of the breast, or other solid tumors curatively treated with no evidence of disease for >3 years, or prostate cancer with a life expectancy of more than 2 years
* Treatment with any approved anticancer agent within last 2 weeks. Any agents must have been stopped at least 2 weeks prior to day 1 of GOAL treatment and all treatment related adverse events must have returned to Grade 1.
* Prior exposition to Obinutuzumab or Pixantrone
* History of hypersensitivity to medicinal products with similar chemical structure as the trial medication
* Active participation in other interventional clinical trials during the present clinical trial or within the last 2 weeks prior to treatment initiation. Concurrent participation in non-treatment studies is not excluded
* Medical or psychological conditions that would jeopardize an adequate and orderly completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Objective overall response rate (ORR) after six treatment cycles or the individual end of treatment | 30 weeks
  The response to treatment is measured by results of computer tomography (CT) for measurable lesions and evaluation for non-measurable lesions after cycle 6 or at the individual end of treatment.

SECONDARY OUTCOMES:
Safety of the combination treatment as measured by the rate of adverse events, which reflects tolerability of the treatment. | 30 weeks
  rate of adverse events
Percentage of patients completing the entire trial treatment | 30 weeks
  Percentage of patients completing the entire trial treatment
Evaluation of best response to trial treatment as measured as best response either during or post the entire treatment | 30 weeks
  best response either during or post the entire treatment
Progression free survival | up to 3 years
  Progression-free survival rate: The time from first intake/dose of trial medication to first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Overall survival | up to 3 years
  * 2-year survival: rate of patients surviving for at least two years after first intake/dose of trial medication.
  * Median overall survival: the time between first applications of trial medication to date of death of half of the patients due to any cause
Overall response rate (ORR) in separate germinal-center B-cell-like (GCB)- vs. non GCB-analysis (gene expression profiling (GEP)) | 30 weeks
  Overall response rate (ORR) in separate germinal-center B-cell-like (GCB)- vs. non GCB-analysis (gene expression profiling (GEP))

CONTACTS AND LOCATIONS:
Overall Officials: Georg Hess, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Department of Hematology, Oncology and Pneumology; University Medical Center of the Johannes Gutenberg-University, Mainz, RLP, Germany